CLINICAL TRIAL: NCT02599649
Title: Phase II Combination of Lirilumab and Nivolumab With 5-Azacitidine in Patients With Myelodysplastic Syndromes (MDS)
Brief Title: Lirilumab and Nivolumab With 5-Azacitidine in Patients With Myelodysplastic Syndromes (MDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment was stopped after the sponsor's decision not to pursue the development of lirilumab for myeloid malignancies.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0934; NCI-2015-02120 (Other: NCI CTRP)
Record Dates: First submitted 2015-11-05; First posted 2015-11-06 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Leukemia
Keywords: Myelodysplastic syndrome; MDS; Low or intermediate-1 MDS; High Risk MDS; Lirilumab; Nivolumab; BMS-936558; Opdivo; Azacitidine; 5-azacytidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Azacytidine
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — lirilumab; Nivolumab; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low or Intermediate-1 MDS Group - Lirilumab (Experimental): Lirilumab by vein over about 60 minutes 1 time each 28 day cycle.
  Interventions: Drug: Lirilumab
- Low or Intermediate-1 MDS Group - Nivolumab + Lirilumab (Experimental): Nivolumab by vein over about 60 minutes every 2 weeks during Cycles 1-9. Lirilumab by vein over about 60 minutes 1 time each cycle. Cycle is 28 days.
  Interventions: Drug: Lirilumab; Drug: Nivolumab
- High Risk MDS Group - Azacitidine + Lirilumab (Experimental): Azacitidine by vein over about 60 minutes on Days 1-7 of each 28 day cycle. Lirilumab by vein over about 60 minutes on Day 7 of each 28 day cycle.
  Interventions: Drug: Lirilumab; Drug: Azacitidine
- High Risk MDS Group - Azacitidine + Lirilumab + Nivolumab (Experimental): Azacitidine by vein over about 60 minutes on Days 1-7 of each 28 day cycle. Lirilumab by vein over about 60 minutes on Day 7 of each 28 day cycle. On Days 7 and 21 of Cycles 1-9 and then on Day 7 of Cycles 10 and beyond, Nivolumab by vein over about 60 minutes.
  Interventions: Drug: Lirilumab; Drug: Nivolumab; Drug: Azacitidine

INTERVENTIONS:
Drug: Lirilumab — 3 mg/kg by vein every 4 weeks.
Drug: Nivolumab — 3 mg/kg by vein on Days 7 and 21 of a 28 day cycle.
  Other Names: BMS-936558; Opdivo
  Arms: High Risk MDS Group - Azacitidine + Lirilumab + Nivolumab; Low or Intermediate-1 MDS Group - Nivolumab + Lirilumab
Drug: Azacitidine — 75 mg/m^2 by vein for 7 days of a 28 day cycle.
  Other Names: 5-azacytidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Azacytidine
  Arms: High Risk MDS Group - Azacitidine + Lirilumab; High Risk MDS Group - Azacitidine + Lirilumab + Nivolumab

SUMMARY:
The goal of this clinical research study is to learn if lirilumab and Opdivo (nivolumab), alone or in combination with Vidaza (azacitidine), can help to control MDS. The safety of these drug combinations will also be studied.

This is an investigational study. Lirilumab is not FDA approved or commercially available. It is currently being used for research purposes. Nivolumab is FDA approved and commercially available for the treatment of melanoma and non small cell lung cancer (NSCLC). Azacitidine is FDA approved and commercially available for the treatment of MDS. The study doctor can explain how the study drugs are designed to work.

Up to 80 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Groups and Study Drug Administration:

If you are found to be eligible to take part in this study, you will be assigned to 1 of 2 study groups based on the status of the disease and then you will be assigned to a cohort based on when you join this study. Each study group will be made up of 2 cohorts. Group 1 is made up of Cohorts A and B. Group 2 is made up of Cohorts C and D. Each cohort will enroll up to 20 participants each.

Each study cycle is 4 weeks.

If you have low risk (low or intermediate-1) MDS, you will be enrolled in Group 1.

* If you are assigned to Cohort A, you will receive lirilumab by vein over about 1 hour 1 time each cycle.
* If you are assigned to Cohort B, you will receive nivolumab by vein over about 1 hour every 2 weeks during Cycles 1-9 and then 1 time each cycle after that. You will also receive lirilumab by vein over about 1 hour 1 time each cycle.

If you have high risk MDS, you will be enrolled in Group 2.

* If you are assigned to Cohort C, you will receive azacitidine by vein for up to 40 minutes on Days 1-7 of each cycle. You will also receive lirilumab by vein over about 1 hour on Day 7 of each cycle.
* If you are assigned to Cohort D, you will receive azacitidine by vein for up to 40 minutes on Days 1-7 of each cycle. You will receive lirilumab by vein over about 1 hour on Day 7 of each cycle. On Days 7 and 21 of Cycles 1-9 and then on Day 7 of Cycles 10 and beyond, you will also receive nivolumab by vein over about 1 hour.

If you are assigned to Cohorts B or D, you will need to stay in the clinic for up to 1 hour after your dose of nivolumab so the study staff may check your vitals and monitor your health for any side effects.

Both you and the study doctor will know to which group you have been assigned.

Study Visits:

One (1) time each week during Cycle 1 and then 1 time during each cycle after that:

* You will have a physical exam.
* Blood (about 2-3 teaspoons) will be drawn for routine tests. These tests may be done more often if your doctor thinks it is needed.

If the doctor thinks it is needed, on Day 28 of Cycle 1 and then every 3 months after that, you will have a bone marrow aspiration to check the status of the disease and for cytogenetic testing.

Every 6 weeks, if you can become pregnant, blood (about 1 teaspoon) or urine will be collected for a pregnancy test.

Length of Study:

You may continue receiving the study drug(s) as long as the study doctor thinks it is in your best interest. You will no longer be able to take the study drug(s) if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

You participation on this study, if you cannot become pregnant, will end after your last dose of study drug(s). If you can become pregnant, your participation on this study will be over after the follow-up pregnancy tests.

Follow-Up Pregnancy Tests:

If you can become pregnant, at 30 days and 70 days after you have stopped taking the study drug(s), blood (about 1 teaspoon) or urine will be collected for a pregnancy test.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with MDS (up to 20% blasts) of any risk. Patients with lower risk MDS (low and int-1 by IPSS) could have received prior non-hypomethylating agent therapy (ie growth factors or lenalidomide). Patients with higher risk MDS (int-2 or high by IPSS) should not have received prior therapy with a hypomethylating agent.
2. Age 18 years or older.
3. Adequate organ function: creatinine </=2.5 x Upper Limit of Normal (ULN); serum bilirubin </=2.5 x ULN; aspartate transaminase (AST) and alanine transaminase (ALT) </=2.5 x ULN.
4. Eastern Cooperative Oncology Group (ECOG) performance status </=2.
5. Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotrophin (beta-hCG) pregnancy test result within 24 hours prior to the first dose of treatment and must agree to use an effective contraception to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug. Females of non- childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy.
6. Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 31 weeks after the last dose of nivolumab.
7. Patients or their legally authorized representative must provide written informed consent.

Exclusion Criteria:

1. History of another primary invasive malignancy that has not been definitively treated or in remission for at least 2 years. Patients with non-melanoma skin cancers or with carcinomas in situ are eligible regardless of the time from diagnosis (including concomitant diagnoses).
2. Any major surgery, radiotherapy, chemotherapy, biologic therapy, immunotherapy, experimental therapy within 2 weeks prior to the first dose of the study drugs.
3. Patients with any other known concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes; cardiovascular disease including congestive heart failure New York Heart Association (NYHA) Class III or IV, myocardial infarction within 6 months, and poorly controlled hypertension; chronic renal failure; or active uncontrolled infection) which, in the opinion of the investigator could compromise participation in the study.
4. Patients unwilling or unable to comply with the protocol.
5. Patients who are on high dose steroid (ie prednisone or equivalent more than 10 mg a day) or immune suppression medications.
6. Patients with autoimmune diseases (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]).
7. Patients with a history of Inflammatory Bowel Disease such as Crohn's disease and ulcerative colitis
8. Patients known to be positive for hepatitis B surface antigen expression or with active hepatitis C infection (positive by polymerase chain reaction or on antiviral therapy for hepatitis C within the last 6 months) or with a history of HIV disease.
9. Current therapy with other systemic anti-neoplastic or anti-neoplastic investigational agents.
10. Females who are pregnant or lactating
11. Prior treatment with stem cell transplantation.
12. Prohibited Prior Treatments and/or Therapies: a) Prior therapy with an anti-KIR, anti-PD-1, or anti-PD-L1, antibody. b) Prior treatment regimens with any immune cell modulating antibody such as anti-CD137 and anti-OX40. However, prior anti-CTLA4 therapy is allowed if the last dose is 101 days or more from the first dose of study drug. c) Exposure to any other investigational drug within 2 weeks prior to the first dose of study drug (within 101 days for anti-CTLA4 therapy). d) Any anti-cancer therapy (e.g., chemotherapy, biologics, vaccines, radiotherapy with curative intent, or hormonal treatment) within 2 weeks prior to the first dose of study drug administration (within 101 days for anti-CTLA4 therapy administration.
13. Continued from #12: e) Use of non-oncology vaccines containing live virus for prevention of infectious diseases within 4 weeks prior to study drug. The use of the inactivated seasonal influenza vaccine (Fluzone®) is allowed. f) Systemic corticosteroid at immunosuppressive doses (> 10 mg/day of prednisone or equivalent), must be discontinued at least 2 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Yalniz FF, Daver N, Rezvani K, Kornblau S, Ohanian M, Borthakur G, DiNardo CD, Konopleva M, Burger J, Gasior Y, Pierce S, Kantarjian H, Garcia-Manero G. A Pilot Trial of Lirilumab With or Without Azacitidine for Patients With Myelodysplastic Syndrome. Clin Lymphoma Myeloma Leuk. 2018 Oct;18(10):658-663.e2. doi: 10.1016/j.clml.2018.06.011. Epub 2018 Jun 15. PMID 30001986
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 2016 to June 2017
Pre-assignment Details: Initially, a sample size of 20 patients for each cohort was planned, but the enrollment was stopped after the sponsor's decision not to pursue the development of lirilumab for myeloid malignancies. The study did not enroll long enough to reach the arms that combined Nivolumab + Lirilumab +/- Azacitidine.
Period: Overall Study
Arm/Group | Low or Intermediate-1 MDS Group - Lirilumab | Low or Intermediate-1 MDS Group - Nivolumab + Lirilumab | High Risk MDS Group - Azacitidine + Lirilumab | High Risk MDS Group - Azacitidine + Lirilumab + Nivolumab
Started | 2 | 0 | 8 | 0
Completed | 2 | 0 | 8 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Initially, a sample size of 20 patients for each cohort was planned, but the enrollment was stopped after the sponsor's decision not to pursue the development of lirilumab for myeloid malignancies. The study did not enroll long enough to reach the arms that combined Nivolumab + Lirilumab +/- Azacitidine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low or Intermediate-1 MDS Group - Lirilumab | Low or Intermediate-1 MDS Group - Nivolumab + Lirilumab | High Risk MDS Group - Azacitidine + Lirilumab | High Risk MDS Group - Azacitidine + Lirilumab + Nivolumab | Total
Number analyzed (Participants) | 2 | 0 | 8 | 0 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0 |  | 0
  Between 18 and 65 years | 0 |  | 3 |  | 3
  >=65 years | 2 |  | 5 |  | 7
Age, Continuous [Median (Full Range); unit: years] | 74 [71 to 76] |  | 70 [50 to 84] |  | 71 [50 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 2 |  | 3
  Male | 1 |  | 6 |  | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 |  | 0
  Asian | 0 |  | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 |  | 0
  Black or African American | 0 |  | 0 |  | 0
  White | 2 |  | 8 |  | 10
  More than one race | 0 |  | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 8 |  | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR) defined as complete response plus partial response (CR + PR) and hematological improvement (HI). MDS International Working Group criteria used to assess response.
Time Frame: 116 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Low or Intermediate-1 MDS Group - Lirilumab | Low or Intermediate-1 MDS Group - Nivolumab + Lirilumab | High Risk MDS Group - Azacitidine + Lirilumab | High Risk MDS Group - Azacitidine + Lirilumab + Nivolumab
Number analyzed (Participants) | 2 | 0 | 8 | 0
Participants | 1 |  | 6 |

ADVERSE EVENTS:
Time Frame: 2 years, 3 months
Description: Initially, a sample size of 20 patients for each cohort was planned, but the enrollment was stopped after the sponsor's decision not to pursue the development of lirilumab for myeloid malignancies. The study did not enroll long enough to reach the arms that combined Nivolumab + Lirilumab +/- Azacitidine.
Arm/Group | Low or Intermediate-1 MDS Group - Lirilumab | Low or Intermediate-1 MDS Group - Nivolumab + Lirilumab | High Risk MDS Group - Azacitidine + Lirilumab | High Risk MDS Group - Azacitidine + Lirilumab + Nivolumab
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0 | 0/8 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/2 | 0/0 | 7/8 | 0/0
Other Adverse Events (participants affected / at risk) | 1/2 | 0/0 | 8/8 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low or Intermediate-1 MDS Group - Lirilumab (N=2) | Low or Intermediate-1 MDS Group - Nivolumab + Lirilumab (N=0) | High Risk MDS Group - Azacitidine + Lirilumab (N=8) | High Risk MDS Group - Azacitidine + Lirilumab + Nivolumab (N=0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Febrile Neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Intracranial Hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small Intestine Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low or Intermediate-1 MDS Group - Lirilumab (N=2) | Low or Intermediate-1 MDS Group - Nivolumab + Lirilumab (N=0) | High Risk MDS Group - Azacitidine + Lirilumab (N=8) | High Risk MDS Group - Azacitidine + Lirilumab + Nivolumab (N=0)
Hyperbilirubinemia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Chest Tightness (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenic Fever (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune Disorder (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Infusion Related Reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT02599649/Prot_SAP_000.pdf